CLINICAL TRIAL: NCT06699875
Title: Comparative Study of the Effectiveness Between Models of Conventional Therapy vs Telerehabilitation With TRAK in Patients Undergoing Axillary Lymph Node Removal (Axillary Lymphadenectomy) as Part of Therapy Against Breast Cancer.
Brief Title: Conventional Therapy vs. Telerehabilitation With TRAK in Patients Undergoing Axillary Lymph Node Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trak Health Solutions S.L. (Industry)
Collaborators: Biogipuzkoa Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAK-LINFA
Record Dates: First submitted 2024-11-14; First posted 2024-11-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; telerehabilitation; telemedicine; digital health; exercise program; physiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The allocation of patients to treatment groups will be performed randomly. IIS Biodonostia will generate the randomization list using R software and enter it into REDCap. This ensures that researchers will neither know nor be able to decide which group each study patient will be randomized to.
  * Control group: The exercise protocol will be completed using printed paper sheets.
  * Treatment group: The exercise protocol is to be completed using the TRAK tool.
Who Masked: Outcomes Assessor
Masking Description: The study will not be blinded to patients because masking the use of an application is impossible. However, mobility assessment will be blinded, so the researchers involved in this task will not know the patient group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAK software intervention group (Experimental): The patients will undergo 4 weeks of treatment using the TRAK platform for shoulder mobility-oriented exercises.
  Interventions: Other: Trak exercise prescription protocol at home
- Paper sheet group (Active Comparator): The patients will undergo 4 weeks of treatment using an exercise paper sheet routine to improve shoulder mobility.
  Interventions: Other: Conventional rehabilitation plan at home

INTERVENTIONS:
Other: Trak exercise prescription protocol at home — Online exercise protocol using the TRAK software. The patient will undergo 4 weeks of an exercise prescription protocol based on shoulder mobility exercises.
  Arms: TRAK software intervention group
Other: Conventional rehabilitation plan at home — Treatment is based on therapeutic exercise following a conventional rehabilitation plan on paper. The patient will undergo 4 weeks of an exercise prescription protocol based on mobility exercises.
  Arms: Paper sheet group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of digital physiotherapy via Trak telerehabilitation with conventional home-based exercises in women who have undergone axillary lymph node removal (axillary lymphadenectomy) as part of breast cancer treatment.

Researchers will compare the Trak telerehabilitation platform to a standard home exercise protocol to assess the impact on shoulder mobility, treatment adherence, and overall patient satisfaction.

Participants will undergo a 4-week home-based rehabilitation using Trak (treatment group) or follow a paper-based exercise protocol (control group) and attend follow-up visits to measure shoulder mobility and any necessary adjustments in treatment.

DETAILED DESCRIPTION:
Women undergoing axillary lymph node removal as part of breast cancer therapy will be recruited. All participants will complete a baseline assessment before being randomly assigned (1:1) to the experimental (telerehabilitation) or control (paper-based exercises) group. Throughout the study, all participants will have follow-up assessments at specific intervals:

* Baseline (V0), initial screening: Health assessments, ensuring their individual needs are met, and written informed consent immediately after the intervention.
* 15 Days Post-Assignment (V1): Initial evaluation of shoulder mobility and assessment for factors like scarring, seroma, and auxiliary cord.
* 3-4 Weeks Post-Assignment (V2): Radiation oncology consultation to assess the mobility metrics and determine whether radiotherapy is necessary or if a delay is required.
* 8 weeks Post-Assessment (V3): The healthcare professional will meet to evaluate shoulder abduction in the affected arm. For patients in the Trak group, the professional will access objective rehabilitation data and metrics from the platform.
* 14 Weeks Post-V1 (V3): Final evaluation of shoulder abduction and assessment of functional recovery (mobility level recovered by the patient). It will also be recorded if the patient needs to receive adjuvant chemotherapy (after surgery). The professional will be able to evaluate each patient's evolution, adherence, and condition. During the visit, the patients will respond to a survey on the technique assigned for rehabilitation (either with the exercises or using Trak).

Patients from the experimental group will use the TRAK telerehabilitation platform (https://www.trakphysio.com/es/) at home for 4 weeks. Patients from the control group will follow a paper-based exercise regimen at home for the same time.

Primary outcomes include shoulder abduction and flexion mobility (first and last visit), adherence to the rehabilitation protocol, satisfaction with the Trak platform (internal survey), and the need for adjuvant chemotherapy. Both groups will complete initial and final assessments on paper, and data will be analyzed for efficacy, adherence, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Female patients equal to or older than 18 years old.
* Patient undergoing axillary lymph node removal (axillary lymphadenectomy) as part of breast cancer therapy.
* Patients with a tablet, smartphone, or laptop who can use electronic devices (or with family support).
* Patient with an e-mail account (or willing to generate a new one).
* Signed the informed consent.

Exclusion Criteria:

* Patient with cognitive restriction
* Patient receiving adjuvant chemotherapy (after lymphadenectomy)
* Patient with previous shoulder-limiting pathology (cuff tear, chronic pain, shoulder fracture with sequelae of limited mobility)
* Patient who has undergone previous surgery on the same shoulder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2023-05-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder abduction mobility | 2-3 days; 15 days; 4-5 and 14 weeks after the surgery
  Active shoulder abduction the patient is able to do actively measurded with a goniometer

SECONDARY OUTCOMES:
Shoulder flexion mobility | 2-3 days; 15 days; 4-5 and 14 weeks after the surgery
  Active shoulder abduction the patient is able to do actively measurded with a goniometer
TRAK designed tool satisfaction questionnaire | 14 weeks
  The trak satisfaction questionnaire was provided to patients in Spanish and consists of 12 questions about usability, usefulness and satisfaction as well as a suggestions section at the end. The score ranges from 0 to 12, with 0 being no satisfaction and 12 being a maximum level of satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Mikel Zabaleta Sistiaga, Principal Investigator — Donostia University Hospital
Locations (1):
- Donostia University Hospital (HU Donostia, OSI Donostialdea), Donostia / San Sebastian, Basque Country, Spain

REFERENCES:
- [Background] Singleton AC, Raeside R, Hyun KK, Partridge SR, Di Tanna GL, Hafiz N, Tu Q, Tat-Ko J, Sum SCM, Sherman KA, Elder E, Redfern J. Electronic Health Interventions for Patients With Breast Cancer: Systematic Review and Meta-Analyses. J Clin Oncol. 2022 Jul 10;40(20):2257-2270. doi: 10.1200/JCO.21.01171. Epub 2022 May 2. PMID 35500200
- [Background] Mahmoud IAM Sr. Usability of Telemedicine in Physical Therapy Rehabilitation: Systematic review. JMIR Rehabil Assist Technol. 2021 Jun 3. doi: 10.2196/25250. Online ahead of print. PMID 34287208
- [Background] Lim JH, Lee HS, Song CS. Home-based rehabilitation programs on postural balance, walking, and quality of life in patients with stroke: A single-blind, randomized controlled trial. Medicine (Baltimore). 2021 Sep 3;100(35):e27154. doi: 10.1097/MD.0000000000027154. PMID 34477171
- [Background] Chae SH, Kim Y, Lee KS, Park HS. Development and Clinical Evaluation of a Web-Based Upper Limb Home Rehabilitation System Using a Smartwatch and Machine Learning Model for Chronic Stroke Survivors: Prospective Comparative Study. JMIR Mhealth Uhealth. 2020 Jul 9;8(7):e17216. doi: 10.2196/17216. PMID 32480361
- [Background] Burns DM, Leung N, Hardisty M, Whyne CM, Henry P, McLachlin S. Shoulder physiotherapy exercise recognition: machine learning the inertial signals from a smartwatch. Physiol Meas. 2018 Jul 23;39(7):075007. doi: 10.1088/1361-6579/aacfd9. PMID 29952759
- [Background] Hosseiniravandi M, Kahlaee AH, Karim H, Ghamkhar L, Safdari R. Home-based telerehabilitation software systems for remote supervising: a systematic review. Int J Technol Assess Health Care. 2020 Apr;36(2):113-125. doi: 10.1017/S0266462320000021. Epub 2020 Mar 10. PMID 32151291
- [Background] Suso-Marti L, La Touche R, Herranz-Gomez A, Angulo-Diaz-Parreno S, Paris-Alemany A, Cuenca-Martinez F. Effectiveness of Telerehabilitation in Physical Therapist Practice: An Umbrella and Mapping Review With Meta-Meta-Analysis. Phys Ther. 2021 May 4;101(5):pzab075. doi: 10.1093/ptj/pzab075. PMID 33611598
- [Background] Sotirova MB, McCaughan EM, Ramsey L, Flannagan C, Kerr DP, O'Connor SR, Blackburn NE, Wilson IM. Acceptability of online exercise-based interventions after breast cancer surgery: systematic review and narrative synthesis. J Cancer Surviv. 2021 Apr;15(2):281-310. doi: 10.1007/s11764-020-00931-6. Epub 2020 Sep 15. PMID 32930924
- [Background] Anton D, Berges I, Bermudez J, Goni A, Illarramendi A. A Telerehabilitation System for the Selection, Evaluation and Remote Management of Therapies. Sensors (Basel). 2018 May 8;18(5):1459. doi: 10.3390/s18051459. PMID 29738442
- [Background] Cramer SC, Dodakian L, Le V, See J, Augsburger R, McKenzie A, Zhou RJ, Chiu NL, Heckhausen J, Cassidy JM, Scacchi W, Smith MT, Barrett AM, Knutson J, Edwards D, Putrino D, Agrawal K, Ngo K, Roth EJ, Tirschwell DL, Woodbury ML, Zafonte R, Zhao W, Spilker J, Wolf SL, Broderick JP, Janis S; National Institutes of Health StrokeNet Telerehab Investigators. Efficacy of Home-Based Telerehabilitation vs In-Clinic Therapy for Adults After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Sep 1;76(9):1079-1087. doi: 10.1001/jamaneurol.2019.1604. PMID 31233135
- [Background] Amin J, Ahmad B, Amin S, Siddiqui AA, Alam MK. Rehabilitation Professional and Patient Satisfaction with Telerehabilitation of Musculoskeletal Disorders: A Systematic Review. Biomed Res Int. 2022 Aug 2;2022:7366063. doi: 10.1155/2022/7366063. eCollection 2022. PMID 35958819
- [Background] Moral-Munoz JA, Zhang W, Cobo MJ, Herrera-Viedma E, Kaber DB. Smartphone-based systems for physical rehabilitation applications: A systematic review. Assist Technol. 2021 Jul 4;33(4):223-236. doi: 10.1080/10400435.2019.1611676. Epub 2019 May 21. PMID 31112461
- [Background] Seron P, Oliveros MJ, Gutierrez-Arias R, Fuentes-Aspe R, Torres-Castro RC, Merino-Osorio C, Nahuelhual P, Inostroza J, Jalil Y, Solano R, Marzuca-Nassr GN, Aguilera-Eguia R, Lavados-Romo P, Soto-Rodriguez FJ, Sabelle C, Villarroel-Silva G, Gomolan P, Huaiquilaf S, Sanchez P. Effectiveness of Telerehabilitation in Physical Therapy: A Rapid Overview. Phys Ther. 2021 Jun 1;101(6):pzab053. doi: 10.1093/ptj/pzab053. PMID 33561280
- [Background] Cheville AL, Moynihan T, Herrin J, Loprinzi C, Kroenke K. Effect of Collaborative Telerehabilitation on Functional Impairment and Pain Among Patients With Advanced-Stage Cancer: A Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):644-652. doi: 10.1001/jamaoncol.2019.0011. PMID 30946436
- [Background] Shenoy P, Shenoy P. Identifying the Challenges and Cost-effectiveness of Telerehabilitation: A Narrative Review. Journal of Clinical and Diagnostic Research. 2018 12;12:1-4
- [Background] Engstrom LO, Oberg B. Patient adherence in an individualized rehabilitation programme: a clinical follow-up. Scand J Public Health. 2005;33(1):11-8. doi: 10.1080/14034940410028299. PMID 15764236
- [Background] Fong SS, Ng SS, Luk WS, Chung JW, Chung LM, Tsang WW, Chow LP. Shoulder Mobility, Muscular Strength, and Quality of Life in Breast Cancer Survivors with and without Tai Chi Qigong Training. Evid Based Complement Alternat Med. 2013;2013:787169. doi: 10.1155/2013/787169. Epub 2013 Apr 23. PMID 23710237
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Servicios | EJIE. (s. f.). Basque Administration Web Portal. Recuperado 27 de octubre de 2022, de https://www.ejie.euskadi.eus/infraestructuras//webejie00-contserv/es/
- [Background] Rees S, Mazuquin B, Richmond H, Williamson E, Bruce J; UK PROSPER Study Group. Role of physiotherapy in supporting recovery from breast cancer treatment: a qualitative study embedded within the UK PROSPER trial. BMJ Open. 2021 May 11;11(5):e040116. doi: 10.1136/bmjopen-2020-040116. PMID 33980512
- [Background] Executive Committee of the International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema: 2020 Consensus Document of the International Society of Lymphology. Lymphology. 2020;53(1):3-19. PMID 32521126
- [Background] Kilbreath SL, Refshauge KM, Beith JM, Ward LC, Lee M, Simpson JM, Hansen R. Upper limb progressive resistance training and stretching exercises following surgery for early breast cancer: a randomized controlled trial. Breast Cancer Res Treat. 2012 Jun;133(2):667-76. doi: 10.1007/s10549-012-1964-1. PMID 22286332
- [Background] Lee TS, Kilbreath SL, Refshauge KM, Herbert RD, Beith JM. Prognosis of the upper limb following surgery and radiation for breast cancer. Breast Cancer Res Treat. 2008 Jul;110(1):19-37. doi: 10.1007/s10549-007-9710-9. Epub 2007 Sep 26. PMID 17899373
- [Background] Ebaugh D, Spinelli B, Schmitz KH. Shoulder impairments and their association with symptomatic rotator cuff disease in breast cancer survivors. Med Hypotheses. 2011 Oct;77(4):481-7. doi: 10.1016/j.mehy.2011.06.015. Epub 2011 Jul 18. PMID 21764521